CLINICAL TRIAL: NCT00227266
Title: Multi-center Phase II Trial of Valproic Acid and Carnitine in Patients With Spinal Muscular Atrophy (SMA CARNI-VAL Trial)
Brief Title: Valproic Acid and Carnitine in Patients With Spinal Muscular Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Families of Spinal Muscular Atrophy (Other); Leadiant Biosciences, Inc. (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13698
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2011-09

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy (SMA); SMA Type 2; SMA Type 3
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Valproic Acid; Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1a (Placebo Comparator): Patients in Cohort 1a - Placebo Comparator, will be on a placebo for 6 months and then will switch to the active treatment. Dosage of the VPA will start at 10-20 mg/kg/day divided into two or tree doses. The dose will be adjusted to achieve a therapeutic trough level of 50-120 micrograms/ml. VPA will be given in the form of 125 mg sprinkle capsules. Dosage for Carnitor will be 50 mg/kg/day with a maximum dose of 10000 mg/day divided into two doses. Carnitor elixir comes as 500 mg/5 ml. All subjects will be given Carnitor or equivalent placebo in the liquid form.
  Interventions: Drug: Valproic Acid and Levocarnitine; Drug: Placebo
- Cohort 1b (Active Comparator): Cohort 1b - Active Comparator will be on treatment throughout the study. Dosage of the VPA will start at 10-20 mg/kg/day divided into two or tree doses. The dose will be adjusted to achieve a therapeutic trough level of 50-120 micrograms/ml. VPA will be given in the form of 125 mg sprinkle capsules. Dosage for Carnitor will be 50 mg/kg/day with a maximum dose of 10000 mg/day divided into two doses. Carnitor elixir comes as 500 mg/5 ml. All subjects will be given Carnitor in the liquid form.
  Interventions: Drug: Valproic Acid and Levocarnitine
- Cohort 2 (Experimental): Cohort 2 pts are on open-label treatment throughout. Dosage of the VPA will start at 10-20 mg/kg/day divided into two or tree doses. The dose will be adjusted to achieve a therapeutic trough level of 50-120 micrograms/ml. VPA will be given in the form of 125 mg sprinkle capsules. Dosage for Carnitor will be 50 mg/kg/day with a maximum dose of 10000 mg/day divided into two doses. Carnitor elixir comes as 500 mg/5 ml. All subjects will be given Carnitor or equivalent placebo in the liquid form.
  Interventions: Drug: Valproic Acid and Levocarnitine

INTERVENTIONS:
Drug: Valproic Acid and Levocarnitine — VPA,sprinkle cap; Levocarnitine, syrup; dosage is by weight
  Other Names: Depakote; VPA; Carnitor
Drug: Placebo
  Arms: Cohort 1a

SUMMARY:
This is a multi-center trial to assess safety and efficacy of a combined regimen of oral valproic acid (VPA) and carnitine in patients with Spinal Muscular Atrophy (SMA) 2 to 17 years of age. Cohort 1 is a double-blind placebo-controlled randomized intention to treat protocol for SMA "sitters" 2 - 8 years of age. Cohort 2 is an open label protocol for SMA "standers and walkers" 3 - 17 years of age to explore responsiveness of efficacy outcomes. Outcome measures will include blood chemistries, functional testing, pulmonary function testing, electrophysiological evaluations, PedsQL quality of life assessment, quantitative assessments of survival motor neuron (SMN) mRNA from blood samples, growth and vital sign parameters. Six centers will enroll a total of 90 patients.

DETAILED DESCRIPTION:
This is a multi-center phase II trial of a combined regimen of oral valproic acid (VPA) and carnitine in patients with Spinal Muscular Atrophy (SMA) 2 to 17 years of age. Cohort 1 is a double-blind placebo-controlled randomized intention to treat protocol for SMA "sitters" 2 - 8 years of age. Subjects will undergo two baseline assessments over 4 to 6 week period, then will be randomized to treatment or placebo for the next six months. All subjects will then be placed on active treatment for the subsequent six month period. Cohort 2 is an open label protocol for SMA "standers and walkers" 3 - 17 years of age to explore responsiveness of efficacy outcomes. Subjects will undergo two baseline assessments over a four to six week period, followed by one year active treatment with VPA and carnitine. Outcome measures are performed every 3 to 6 months, and include blood chemistries, functional testing, pulmonary function testing, electrophysiological evaluations, PedsQL quality of life assessment, quantitative assessments of survival motor neuron (SMN) mRNA from blood samples, growth and vital sign parameters. Six centers will enroll a total of 90 patients.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* Confirmed genetic diagnosis of 5q SMA
* SMA 2 or non-ambulatory SMA 3: all subjects must be able to sit independently for at least 3 seconds without support
* Age 2 to 8 years at time of enrollment

Cohort 2

* Confirmed genetic diagnosis of 5q SMA
* SMA subjects (SMA types 2 or 3) who can stand independently without braces or other support for up to 2 seconds, or walk independently
* Age 3 to 17 years at time of study enrollment

Exclusion Criteria:

Cohort 1

* Need for BiPAP support > 12 hours per day
* Spinal rod or fixation for scoliosis or anticipated need within six months of enrollment
* Inability to meet study visit requirements or cooperate reliably with functional testing
* Coexisting medical conditions that contraindicate travel, testing or study medications
* Use of medications or supplements which interfere with valproic acid or carnitine metabolism within 3 months of study enrollment.
* Current use of either VPA or carnitine. If study subject is taking VPA or carnitine then patient must go through a washout period of 12 weeks before enrollment into the study
* Body Mass Index > 90th % for age

Cohort 2

* Spinal rod or fixation for scoliosis or anticipated need within six months of enrollment
* Inability to meet study visit requirements or cooperate with functional testing
* Transaminases, amylase or lipase > 3.0 x normal values, WBC < 3.0 or neutropenia < 1.0, platelets < 100 K, or hematocrit < 30 persisting over a 30 day period.
* Coexisting medical conditions that contraindicate travel, testing or study medications
* Use of medications or supplements which interfere with valproic acid or carnitine metabolism within 3 months of study enrollment.
* Current use of either VPA or carnitine. If study subject is taking VPA or carnitine then patient must be go through a washout period of 12 weeks before enrollment in the study.
* Body Mass Index > 90th % for age
* Pregnant women/girls, or those intending to try to become pregnant during the course of the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2005-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn J Swoboda, M.D., Principal Investigator — University of Utah/Primary Children's Medical Center
Locations (6):
- United States (5):
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Ohio State University, Columbus, Ohio
  - University of Utah/Primary Children's Medical Center, Salt Lake City, Utah
  - University of Wisconsin Children's Hospital, Madison, Wisconsin
- Hospital Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Background] Brahe C, Bertini E. Spinal muscular atrophies: recent insights and impact on molecular diagnosis. J Mol Med (Berl). 1996 Oct;74(10):555-62. doi: 10.1007/s001090050059. PMID 8912176
- [Background] Roberts DF, Chavez J, Court SD. The genetic component in child mortality. Arch Dis Child. 1970 Feb;45(239):33-8. doi: 10.1136/adc.45.239.33. PMID 4245389
- [Background] Pearn J. Incidence, prevalence, and gene frequency studies of chronic childhood spinal muscular atrophy. J Med Genet. 1978 Dec;15(6):409-13. doi: 10.1136/jmg.15.6.409. PMID 745211
- [Background] Czeizel A, Hamula J. A hungarian study on Werdnig-Hoffmann disease. J Med Genet. 1989 Dec;26(12):761-3. doi: 10.1136/jmg.26.12.761. PMID 2614795
- [Background] Emery AE. Population frequencies of inherited neuromuscular diseases--a world survey. Neuromuscul Disord. 1991;1(1):19-29. doi: 10.1016/0960-8966(91)90039-u. PMID 1822774
- [Background] Merlini L, Stagni SB, Marri E, Granata C. Epidemiology of neuromuscular disorders in the under-20 population in Bologna Province, Italy. Neuromuscul Disord. 1992;2(3):197-200. doi: 10.1016/0960-8966(92)90006-r. PMID 1483045
- [Background] Pearn J. Classification of spinal muscular atrophies. Lancet. 1980 Apr 26;1(8174):919-22. doi: 10.1016/s0140-6736(80)90847-8. PMID 6103267
- [Background] Bromberg MB, Swoboda KJ. Motor unit number estimation in infants and children with spinal muscular atrophy. Muscle Nerve. 2002 Mar;25(3):445-7. doi: 10.1002/mus.10050. PMID 11870724
- [Background] Swoboda KJ, Prior TW, Scott CB, McNaught TP, Wride MC, Reyna SP, Bromberg MB. Natural history of denervation in SMA: relation to age, SMN2 copy number, and function. Ann Neurol. 2005 May;57(5):704-12. doi: 10.1002/ana.20473. PMID 15852397
- [Background] Crawford TO. From enigmatic to problematic: the new molecular genetics of childhood spinal muscular atrophy. Neurology. 1996 Feb;46(2):335-40. doi: 10.1212/wnl.46.2.335. No abstract available. PMID 8614490
- [Background] Gilliam TC, Brzustowicz LM, Castilla LH, Lehner T, Penchaszadeh GK, Daniels RJ, Byth BC, Knowles J, Hislop JE, Shapira Y, et al. Genetic homogeneity between acute and chronic forms of spinal muscular atrophy. Nature. 1990 Jun 28;345(6278):823-5. doi: 10.1038/345823a0. PMID 1972783
- [Background] Melki J, Lefebvre S, Burglen L, Burlet P, Clermont O, Millasseau P, Reboullet S, Benichou B, Zeviani M, Le Paslier D, et al. De novo and inherited deletions of the 5q13 region in spinal muscular atrophies. Science. 1994 Jun 3;264(5164):1474-7. doi: 10.1126/science.7910982.
- [Background] Monani UR, Lorson CL, Parsons DW, Prior TW, Androphy EJ, Burghes AH, McPherson JD. A single nucleotide difference that alters splicing patterns distinguishes the SMA gene SMN1 from the copy gene SMN2. Hum Mol Genet. 1999 Jul;8(7):1177-83. doi: 10.1093/hmg/8.7.1177. PMID 10369862
- [Background] Campbell L, Potter A, Ignatius J, Dubowitz V, Davies K. Genomic variation and gene conversion in spinal muscular atrophy: implications for disease process and clinical phenotype. Am J Hum Genet. 1997 Jul;61(1):40-50. doi: 10.1086/513886. PMID 9245983
- [Background] Lefebvre S, Burlet P, Liu Q, Bertrandy S, Clermont O, Munnich A, Dreyfuss G, Melki J. Correlation between severity and SMN protein level in spinal muscular atrophy. Nat Genet. 1997 Jul;16(3):265-9. doi: 10.1038/ng0797-265. PMID 9207792
- [Background] Monani UR, Sendtner M, Coovert DD, Parsons DW, Andreassi C, Le TT, Jablonka S, Schrank B, Rossoll W, Prior TW, Morris GE, Burghes AH. The human centromeric survival motor neuron gene (SMN2) rescues embryonic lethality in Smn(-/-) mice and results in a mouse with spinal muscular atrophy. Hum Mol Genet. 2000 Feb 12;9(3):333-9. doi: 10.1093/hmg/9.3.333. PMID 10655541
- [Background] Feldkotter M, Schwarzer V, Wirth R, Wienker TF, Wirth B. Quantitative analyses of SMN1 and SMN2 based on real-time lightCycler PCR: fast and highly reliable carrier testing and prediction of severity of spinal muscular atrophy. Am J Hum Genet. 2002 Feb;70(2):358-68. doi: 10.1086/338627. Epub 2001 Dec 21. PMID 11791208
- [Background] Mailman MD, Heinz JW, Papp AC, Snyder PJ, Sedra MS, Wirth B, Burghes AH, Prior TW. Molecular analysis of spinal muscular atrophy and modification of the phenotype by SMN2. Genet Med. 2002 Jan-Feb;4(1):20-6. doi: 10.1097/00125817-200201000-00004. PMID 11839954
- [Background] Fischer U, Liu Q, Dreyfuss G. The SMN-SIP1 complex has an essential role in spliceosomal snRNP biogenesis. Cell. 1997 Sep 19;90(6):1023-9. doi: 10.1016/s0092-8674(00)80368-2. PMID 9323130
- [Background] Chang JG, Hsieh-Li HM, Jong YJ, Wang NM, Tsai CH, Li H. Treatment of spinal muscular atrophy by sodium butyrate. Proc Natl Acad Sci U S A. 2001 Aug 14;98(17):9808-13. doi: 10.1073/pnas.171105098. PMID 11504946
- [Background] Andreassi C, Jarecki J, Zhou J, Coovert DD, Monani UR, Chen X, Whitney M, Pollok B, Zhang M, Androphy E, Burghes AH. Aclarubicin treatment restores SMN levels to cells derived from type I spinal muscular atrophy patients. Hum Mol Genet. 2001 Nov 15;10(24):2841-9. doi: 10.1093/hmg/10.24.2841. PMID 11734549
- [Background] Brichta L, Hofmann Y, Hahnen E, Siebzehnrubl FA, Raschke H, Blumcke I, Eyupoglu IY, Wirth B. Valproic acid increases the SMN2 protein level: a well-known drug as a potential therapy for spinal muscular atrophy. Hum Mol Genet. 2003 Oct 1;12(19):2481-9. doi: 10.1093/hmg/ddg256. Epub 2003 Jul 29. PMID 12915451
- [Background] Andreassi C, Angelozzi C, Tiziano FD, Vitali T, De Vincenzi E, Boninsegna A, Villanova M, Bertini E, Pini A, Neri G, Brahe C. Phenylbutyrate increases SMN expression in vitro: relevance for treatment of spinal muscular atrophy. Eur J Hum Genet. 2004 Jan;12(1):59-65. doi: 10.1038/sj.ejhg.5201102. PMID 14560316
- [Background] Bohmer T, Rydning A, Solberg HE. Carnitine levels in human serum in health and disease. Clin Chim Acta. 1974 Nov 20;57(1):55-61. doi: 10.1016/0009-8981(74)90177-6. No abstract available. PMID 4279150
- [Background] Brooks H, Goldberg L, Holland R, Klein M, Sanzari N, DeFelice S. Carnitine-induced effects on cardiac and peripheral hemodynamics. J Clin Pharmacol. 1977 Oct;17(10 Pt 1):561-8. doi: 10.1177/009127007701701003. No abstract available. PMID 915022
- [Background] Christiansen RZ, Bremer J. Active transport of butyrobetaine and carnitine into isolated liver cells. Biochim Biophys Acta. 1976 Nov 2;448(4):562-77. doi: 10.1016/0005-2736(76)90110-3. PMID 974147
- [Background] Lindstedt S, Lindstedt G. Distribution and Excretion of Carnitine in the Rat. Acta. Chem. Scand. 1961;15:701-702
- [Background] Rebouche CJ, Engel AG. Carnitine metabolism and deficiency syndromes. Mayo Clin Proc. 1983 Aug;58(8):533-40. PMID 6348429
- [Background] Rebouche CJ, Paulson DJ. Carnitine metabolism and function in humans. Annu Rev Nutr. 1986;6:41-66. doi: 10.1146/annurev.nu.06.070186.000353. PMID 3524622
- [Background] Igarashi N, Sato T, Kyouya S. Secondary carnitine deficiency in handicapped patients receiving valproic acid and/or elemental diet. Acta Paediatr Jpn. 1990 Apr;32(2):139-45. doi: 10.1111/j.1442-200x.1990.tb00799.x. PMID 2143048
- [Background] Thurston JH, Hauhart RE. Amelioration of adverse effects of valproic acid on ketogenesis and liver coenzyme A metabolism by cotreatment with pantothenate and carnitine in developing mice: possible clinical significance. Pediatr Res. 1992 Apr;31(4 Pt 1):419-23. doi: 10.1203/00006450-199204000-00023. PMID 1570210
- [Background] Tein I, DiMauro S, Xie ZW, De Vivo DC. Valproic acid impairs carnitine uptake in cultured human skin fibroblasts. An in vitro model for the pathogenesis of valproic acid-associated carnitine deficiency. Pediatr Res. 1993 Sep;34(3):281-7. doi: 10.1203/00006450-199309000-00008. PMID 8134167
- [Background] Melegh B, Pap M, Morava E, Molnar D, Dani M, Kurucz J. Carnitine-dependent changes of metabolic fuel consumption during long-term treatment with valproic acid. J Pediatr. 1994 Aug;125(2):317-21. doi: 10.1016/s0022-3476(94)70218-7. PMID 8040784
- [Background] Tein I, Xie ZW. Reversal of valproic acid-associated impairment of carnitine uptake in cultured human skin fibroblasts. Biochem Biophys Res Commun. 1994 Oct 28;204(2):753-8. doi: 10.1006/bbrc.1994.2523. PMID 7980539
- [Background] Van Wouwe JP. Carnitine deficiency during valproic acid treatment. Int J Vitam Nutr Res. 1995;65(3):211-4. PMID 8830002
- [Background] Evangeliou A, Vlassopoulos D. Carnitine metabolism and deficit--when supplementation is necessary? Curr Pharm Biotechnol. 2003 Jun;4(3):211-9. doi: 10.2174/1389201033489829. PMID 12769764
- [Background] Coulter DL. Carnitine deficiency: a possible mechanism for valproate hepatotoxicity. Lancet. 1984 Mar 24;1(8378):689. doi: 10.1016/s0140-6736(84)92209-8. No abstract available. PMID 6142383
- [Background] Coulter DL. Carnitine, valproate, and toxicity. J Child Neurol. 1991 Jan;6(1):7-14. doi: 10.1177/088307389100600102. PMID 2002205
- [Background] Scriver C, Beautet A, Sly W, Valle D. The Metabolic Basis of Inherited Disease. New York: McGraw Hill, 1989
- [Background] Schaub J, Van Hoof F, Vis H. Inborn Errors of Metabolism. New York: Raven Press, 1991
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Derived] Kissel JT, Scott CB, Reyna SP, Crawford TO, Simard LR, Krosschell KJ, Acsadi G, Elsheik B, Schroth MK, D'Anjou G, LaSalle B, Prior TW, Sorenson S, Maczulski JA, Bromberg MB, Chan GM, Swoboda KJ; Project Cure Spinal Muscular Atrophy Investigators' Network. SMA CARNIVAL TRIAL PART II: a prospective, single-armed trial of L-carnitine and valproic acid in ambulatory children with spinal muscular atrophy. PLoS One. 2011;6(7):e21296. doi: 10.1371/journal.pone.0021296. Epub 2011 Jul 6. PMID 21754985
- [Derived] Swoboda KJ, Scott CB, Crawford TO, Simard LR, Reyna SP, Krosschell KJ, Acsadi G, Elsheik B, Schroth MK, D'Anjou G, LaSalle B, Prior TW, Sorenson SL, Maczulski JA, Bromberg MB, Chan GM, Kissel JT; Project Cure Spinal Muscular Atrophy Investigators Network. SMA CARNI-VAL trial part I: double-blind, randomized, placebo-controlled trial of L-carnitine and valproic acid in spinal muscular atrophy. PLoS One. 2010 Aug 19;5(8):e12140. doi: 10.1371/journal.pone.0012140. PMID 20808854

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject's were recruited during the periods of September 2005 to September 2006 across the United States.
Groups:
- Cohort 1a Sitters Placebo Then Treatment: Dosage of the VPA will start at 10-20 mg/kg/day divided into two or tree doses. The dose will be adjusted to achieve a therapeutic trough level of 50-120 micrograms/ml. VPA will be given in the form of 125 mg sprinkle capsules. Dosage for Carnitor will be 50 mg/kg/day with a maximum dose of 10000 mg/day divided into two doses. Carnitor elixir comes as 500 mg/5 ml. All subjects will be given Carnitor or equivalent placebo in the liquid form.
- Cohort 1b Sitters Treatment; Cohort 2 Standers and Walkers - Treatment: Dosage of the VPA will start at 10-20 mg/kg/day divided into two or tree doses. The dose will be adjusted to achieve a therapeutic trough level of 50-120 micrograms/ml. VPA will be given in the form of 125 mg sprinkle capsules. Dosage for Carnitor will be 50 mg/kg/day with a maximum dose of 10000 mg/day divided into two doses. Carnitor elixir comes as 500 mg/5 ml. All subjects will be given Carnitor in the liquid form.
Period: Overall Study
Arm/Group | Cohort 1a Sitters Placebo Then Treatment | Cohort 1b Sitters Treatment | Cohort 2 Standers and Walkers - Treatment
Started | 31 | 30 | 33
Completed | 30 | 30 | 29
Not Completed | 1 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Excessive weight gain | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a Sitters Placebo Then Treatment | Cohort 1b Sitters Treatment | Cohort 2 Standers and Walkers - Treatment | Total
Number analyzed (Participants) | 31 | 30 | 33 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 30 | 33 | 94
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.4 (1.9) | 4.3 (2.1) | 7.3 (3.7) | 5.4 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 11 | 39
  Male | 20 | 13 | 22 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 29 | 27 | 30 | 86
  Unknown or Not Reported | 0 | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 26 | 25 | 29 | 80
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 29 | 80
  Canada | 6 | 4 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety Labs
Description: Participants will have labs drawn regularly to maintain appropriate dosing and monitor liver function
Time Frame: -4 wks, 0, 2 wks, 3 mo, 6 mo, 9 mo, 12 mo for safety labs; throughout for AEs
Reporting Status: Not Posted

2. Primary Outcome: Efficacy, Measured Through Motor Function Assessments
Time Frame: -4wks, 0, 3 mo, 6 mo, 12 mo
Reporting Status: Not Posted

3. Secondary Outcome: Quantitative Assessment of SMN mRNA From Blood Samples
Time Frame: -4wks or 0, 3 mo, 6 mo, 12 mo
Reporting Status: Not Posted

4. Secondary Outcome: Peds QL™ Assessment: Parental Version (All), Child Versions (> 5yrs)
Time Frame: -4wks, 0, 3mo, 6mo, 12mo
Reporting Status: Not Posted

5. Secondary Outcome: Max CMAP Amplitude (Mean)
Description: The maximum Compound Motor Action Potential (CMAP) is a measurement obtained through EMG testing that is associated with disease progression. In this study, we measure the maximum CMAP by stimulating one nerve in the hand and measuring the response of the muscle. This is done multiple times, the outcome used is the highest peak, or response observed.
Time Frame: 1 month prior to official enrollment, beginning of study (0 months), 6 months, 12 months (data point not available)
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Cohort 1a Sitters Placebo Then Treatment | Cohort 1b Sitters Treatment | Cohort 2 Standers and Walkers - Treatment
Number analyzed (Participants) | 23 | 21 | 24
mV
  Baseline | 2.28 (1.55) | 2.93 (1.56) | 5.52 (2.56)
  6 months | 2.32 (1.75) | 2.37 (1.82) | 6.56 (2.99)

6. Secondary Outcome: Max CMAP Amplitude Median
Description: as for outcome 5
Time Frame: 1 month prior to official enrollment, beginning of study (0 months), 6 months, 12 months (data point not available)
Measure: Median (Full Range); unit: mV
Arm/Group | Cohort 1a Sitters Placebo Then Treatment | Cohort 1b Sitters Treatment | Cohort 2 Standers and Walkers - Treatment
Number analyzed (Participants) | 23 | 21 | 24
mV
  Baseline | 1.91 [0.5 to 7.66] | 2.2 [0.5 to 6.66] | 5.3 [1.2 to 10.42]
  6 months | 1.44 [0.5 to 6.14] | 1.8 [0.3 to 7.81] | 5.85 [1.50 to 12.20]

7. Secondary Outcome: Ulnar MUNE
Time Frame: -4 wks, 0, 3 mo, 6 mo, 12 mo
Reporting Status: Not Posted

8. Secondary Outcome: Growth and Vital Sign Parameters
Time Frame: -4 wks, 0, 3mo, 6mo, 12mo
Reporting Status: Not Posted

9. Secondary Outcome: Nutritional Status
Time Frame: -4 wks, 0, 3mo, 6mo, 12mo
Reporting Status: Not Posted

10. Post Hoc Outcome: Modified Hammersmith Extend Baseline
Description: Baseline Modified Hammersmith Extend testing. The baseline test is the score they receive during their screening visits. This scale ranges from 0 to 56. A higher score indicates a better outcome.
  This scale is used to assess gross motor abilities of children with SMA in multiple research trials as well as in clinical settings.
Time Frame: 1 month prior to enrollment, at enrollment (0 months)
Population: Analysis was determined per protocol
Measure: Mean (Full Range); unit: Score
Groups:
- Cohort 2 Experimental: Patients in cohort 2 (SMA "standers and walkers") will receive VPA + Carnitine treatment for the entire 12 month time period.
Arm/Group | Cohort 2 Experimental
Number analyzed (Participants) | 33
Score
  Modified Hammersmith Extend at S1 (-4 weeks) | 47.0 [29 to 56]
  Modified Hammersmith Extend at S2 (0 weeks) | 48.3 [36 to 56]
Statistical Analysis 1: Comparison: Cohort 2 Experimental; MHFMS-Extend was not normally distributed at p=0.048. Test-retest reliability of MHFMS-Extend measurements from the first (S1) to the second (S2) screening visit was analyzed using Spearman's correlation; Test type: Superiority or Other; p < 0.001, Spearman's correlation; Spearman's correlation = 0.93

11. Primary Outcome: Modified Hammersmith Change From Baseline to 6 Months
Description: Comparison of Modified Hammersmith Change from baseline to 6 months. Scores range from 0 to 40. A higher score indicates a better outcome. This scale is used to assess gross motor abilities of non-ambulant children with SMA in multiple research trials as well as in clinical settings.
Time Frame: 0 months, 6 months
Population: Analysis only pertains to cohort 1a and 1b.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Cohort 1a Sitters Placebo Then Treatment | Cohort 1b Sitters Treatment
Number analyzed (Participants) | 31 | 30
Score
  Baseline visit (0 weeks) | 20.0 (9.3) | 16.6 (8.7)
  6 Month visit (V2) | 20.6 (8.1) | 16.8 (7.9)
  Change from Baseline | 0.6 (3.98) | 0.2 (2.88)

12. Secondary Outcome: DEXA
Time Frame: 0, 6mo, 12mo
Reporting Status: Not Posted

13. Secondary Outcome: Max CMAP Area (Mean)
Description: The maximum Compound Motor Action Potential (CMAP) area is a measurement obtained through EMG testing that is associated with disease progression. In this study, we measure the maximum CMAP by stimulating one nerve in the hand and measuring the response of the muscle. This procedure is repeated multiple times. The maximum area is the response that results in the largest area under the response curve.
Time Frame: 1 month prior to official enrollment, beginning of study (0 months), 6 months, 12 months (data point not available)
Measure: Mean (Standard Deviation); unit: mVms
Arm/Group | Cohort 1a Sitters Placebo Then Treatment | Cohort 1b Sitters Treatment | Cohort 2 Standers and Walkers - Treatment
Number analyzed (Participants) | 23 | 21 | 24
mVms
  Baseline | 5.46 (5.03) | 5.45 (4.23) | 14.85 (7.68)
  6 months | 5.28 (4.49) | 5.26 (4.65) | 16.26 (7.13)

14. Secondary Outcome: Max CMAP Area (Median)
Description: as for outcome 13
Time Frame: 1 month prior to official enrollment, beginning of study (0 months), 6 months, 12 months (data point not available)
Measure: Median (Full Range); unit: mVms
Arm/Group | Cohort 1a Sitters Placebo Then Treatment | Cohort 1b Sitters Treatment | Cohort 2 Standers and Walkers - Treatment
Number analyzed (Participants) | 23 | 21 | 24
mVms
  Baseline | 3.6 [0.7 to 19.71] | 4.6 [1.3 to 16.78] | 13.65 [2.6 to 38.29]
  6 months | 3.74 [0.6 to 16.13] | 3.4 [0.6 to 18.81] | 16.85 [3.7 to 29.10]

ADVERSE EVENTS:
Time Frame: Phase 1 Serious Adverse Events (time period during which placebo (1a) and treatment (1b)were randomly treated): 6 months. And Phase 1 and 2 Adverse Events: 12 months
Arm/Group | Cohort 1a Sitters Placebo Then Treatment | Cohort 1b Sitters Treatment | Cohort 2 Standers and Walkers - Treatment
Serious Adverse Events (participants affected / at risk) | 1/31 | 4/30 | 4/33
Other Adverse Events (participants affected / at risk) | 18/31 | 23/30 | 28/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a Sitters Placebo Then Treatment (N=31) | Cohort 1b Sitters Treatment (N=30) | Cohort 2 Standers and Walkers - Treatment (N=33)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
General Disorder (General disorders) | 0 | 1 | 0 — Pyrexia
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pneumonitis (Infections and infestations) | 0 | 1 | 0
Skin Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tachyponea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a Sitters Placebo Then Treatment (N=31) | Cohort 1b Sitters Treatment (N=30) | Cohort 2 Standers and Walkers - Treatment (N=33)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 3 | 7
Agitation (Nervous system disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Chocking Sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 4
Croup (Infections and infestations) | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Dermatitis Allergic (Immune system disorders) | 3 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Ear Infection (Infections and infestations) | 2 | 3 | 4
Emotional Disorder of Childhood (Psychiatric disorders) | 2 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1
Femur Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Forearm Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gastroesophagheal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Hand Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Impulsive Behaviour (Nervous system disorders) | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Increased Urination Frequency (Renal and urinary disorders) | 1 | 0 | 0
Irritability (Nervous system disorders) | 2 | 1 | 0
Join Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0
Multiple Allergies (Immune system disorders) | 0 | 2 | 5
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 2
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Patella Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Pharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2
Pneumonitis (Infections and infestations) | 1 | 1 | 0
Pyrexia (General disorders) | 4 | 5 | 7
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tinea Infection (Infections and infestations) | 0 | 1 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 6 | 12 | 6
Weight Incresed (Investigations) | 4 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No